CLINICAL TRIAL: NCT00500773
Title: Investigation of Myocardial Injury, Ventricular Dysfunction and Cardiovascular Risk Factors in Different Groups of Marathon Runners
Brief Title: Investigation of Cardiac Function and Cardiovascular Risk Factors in Marathon Runners- The Munich Marathon Study
Acronym: MMS
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Dr. med. Henner Hanssen, Lehrstuzl für Praeventive und rehabilitative Sportmedizin
Other Study IDs: 1807/07
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Modes of Exercise and Myocardial and Endothelial Function; Microcirculation; Subclinical Endorgan Damage; Obesity
Keywords: cardiovascular risc factors; inflammation; aerobic and exertional exercise
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the cardiovascular risk involved in the exertional exercise of marathon running. The researchers aim to investigate the beneficial effects of regular well-dosed exercise on health and compare these findings with the effects of the extreme strains of marathon running. Subclinical injuries to heart and arteries are being investigated in different groups of runners, including obese participants.

DETAILED DESCRIPTION:
Regular exercise leads to an improvement of cardiovascular risc factors in patients with coronary heart disease, atherosclerosis and metabolic disorders. Aerobic exercise has anti-inflammatory effects. In contrast, the exertional exercise of marathon running causes an acute pro-inflammatory impulse. This may lead to myocardial injury and, in case of preexisting plaques, may result in plaque rupture and acute myocardial infarction.

The researchers aim to define the critical role of inflammatory markers and cardiovascular risk factors as a predictor of an increased risk for myocardial and endothelial dysfunction in marathon runners.

The study groups are divided into average trained runners (40 km/week), average trained obese runners and highly trained runners (> 70km/week). Training programmes are supervised by professional coaches. Individual scientific marathon contests are organized for the assessments.

Diagnostic tools include measurements of pulse wave velocity and heart rate turbulence, echocardiography and, for the first time, MRI-scans pre- and post marathon running. Additionally, cardiovascular markers such as endothelial progenitor cells (EPCs)and adiponectin are measured. Inflammatory markers include c-reactive protein (CRP), interleukins and tumor necrosis factor.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 30-60 years
* Obese subjects: BMI > 27 and waist circumference > 102cm

Exclusion Criteria:

* manifested heart disease
* insulin dependent diabetes mellitus
* multiple drug therapy
* GFR < 60 ml/min.
* claustrophobia
* metal implants

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male marathon runners with no more than one treated cardiovascular risk factor aged 30-60 years. Participation of at least a 1/2 marathon in recent history.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henner Hanssen, MD, Principal Investigator — Department of Prevention and Sportmedicine, Technical University Munich
Locations (1):
- Department of Prevention and Sportsmedicine, Technical University of Munich, Connollystrasse 32, Munich, Bavaria, Germany

REFERENCES:
- See also: Institutional homepage — http://www.sport.med.tum.de